CLINICAL TRIAL: NCT01376752
Title: A Phase III Randomized Study Evaluating Hyperthermic Intra-Peritoneal Chemotherapy (HIPEC) in the Treatment of Relapse Ovarian Cancer
Brief Title: Hyperthermic Intra-Peritoneal Chemotherapy (HIPEC) in Relapse Ovarian Cancer Treatment
Acronym: CHIPOR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FEDEGYN 02 / 0410-CHIPOR; 2010-023035-42 (EudraCT Number)
Record Dates: First submitted 2011-03-28; First posted 2011-06-20 (Estimated); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Epithelial Cancer Recurrent
MeSH Terms: interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- maximal cytoreductive surgery without HIPEC (Active Comparator): The participant will have a regular cytoreductive surgery without the adjunction of HIPEC.
  Interventions: Procedure: Maximal cytoreductive surgery
- maximal cytoreductive surgery with HIPEC (Experimental): The participant will have a regular cytoreductive surgery, then the adjunction of HIPEC: hyperthermic cisplatin will be used at 75mg/m²
  Interventions: Procedure: Maximal cytoreductive surgery; Drug: HIPEC

INTERVENTIONS:
Procedure: Maximal cytoreductive surgery — Maximal cytoreductive surgery
Drug: HIPEC — HIPEC: Hyperthermic Intra-PEritoneal Chemotherapy. Administration of cisplatin at 75mg/m²
  Arms: maximal cytoreductive surgery with HIPEC

SUMMARY:
CHIPOR hypothesis is that the adjunction of platinum HIPEC in first relapsed epithelial ovarian cancer is able to improve the median Overall Survival (OS) by 12 months. In that hypothesis, with alpha risk of 5%, a power beta of 80%, during a 3 years period of inclusion and a 3 years follow-up, the number of patients to include is 404. Taking into account a 10% failure, an overall number of 444 patients is required.

DETAILED DESCRIPTION:
The patient received before the surgery a second line chemotherapy, platinum-based regimen with either carboplatine-paclitaxel, or carboplatine-caelyx. At the end of the six courses IV chemotherapy, if the disease is still responding and if a complete cytoreductive surgery seems possible, the patient is included after signed informed consent and will be operated 5 to 8 weeks after the last second-line chemotherapy cycle.

So, during the surgery the patient will be randomized if the complete cytoreductive surgery is really done and will then receive:

* either treatment A = maximal cytoreductive surgery without HIPEC
* or treatment B = maximal cytoreductive surgery with HIPEC

The HIPEC will be done at the end of the surgery. At the end of cytoreductive surgery, tumor residual disease must be null or very limited (Sugarbaker completeness cytoreduction: CC0 (no residual)-CC1 (residual < 0.25cm).

Two methods will be used for the HIPEC: Open or closed abdomen, depends on the site practice. Each site will use the same method during the study for all included patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years
* Performance Status WHO < 2
* Initially treated for Epithelial Ovarian Carcinoma
* Patient with only peritoneal relapse occurred at least 6 month from the initial treatment, resectable without distant metastasis (with the exception of communicating pleura effusion, sensitive to platine-based second line chemotherapy and resectable lymph-nodes in the groin or retro peritoneal)
* Platinum based second-line chemotherapy before surgery with either carboplatine-paclitaxel, or carboplatine-caelyx
* Complete cytoreductive surgery
* The surgery has to be planned 5 to 8 weeks from the last 2nd of chemotherapy
* No hepatic failure, bilirubin ≤ 1,5 time the Normal limit, ASAT and ALAT ≤ 3 time the Upper Normal Limit
* No Renal insufficiency (serum creatinine < 1,5 time the normal limit, creatinine clearance > 80 mL/min). calculated with MDRD method
* Hematology function: PNN ≥ 1,5x10⁹/L, platelets ≥ 100x10⁹/L
* No contraindication to general anaesthesia for heavy surgery
* Patients having read, signed and dated Informed consent before any study procedure
* Childbearing patients have to take appropriate contraceptive methods during the treatment and until 6 months after the treatment

Exclusion Criteria:

* Patient age <18 years
* Previous cancer in the last 5 years (except cutaneous baso-cellular epithelioma or uterine peripheral epithelioma)
* Hypersensitivity to Platinum compound
* Distant metastasis
* Use of anti-angiogenic treatment
* Patient with other concurrent severe life threatening disease
* The need to perform more than two segmental digestive resections during the CRS +/- HIPEC surgery
* Any progressive disease during the IV systemic second-line chemotherapy (platine-based)
* Incomplete cytoreductive surgery with macroscopical residual disease (Sugarbaker > CC1)
* Early relapse: less than 6 mois after the end of the first treatment
* Ovarian tumor other than Epithelioma Ovarian Cancer
* Uncontrolled infection
* Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Clinically significant cardiovascular disease contraindicating the hyper hydratation, which is necessary for HIPEC
* Patient already treated with HIPEC for the ovarian cancer
* Individual deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2011-04-26 (Actual); Primary Completion 2023-01-08 (Actual); Study Completion 2027-05-14 (Estimated)

PRIMARY OUTCOMES:
overall survival | from randomization to death (up to 4 years)
  Follow-up of 4 years.

SECONDARY OUTCOMES:
relapse free survival | from randomization to relapse (up to 4 years)
  Follow-up of 4 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc CLASSE, Principal Investigator — Centre rené Gauducheau, NANTES
Locations (33):
- Institut Jules Bordet, Brussels, Belgium
- France (31):
  - CHU d'AMIENS, Amiens
  - Centre Paul Papin, Angers
  - Institut Bergonie, Bordeaux
  - Clinique Pasteur, Brest
  - Polyclinique Kéraudren, Brest
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre hospitalier de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - Clinique Victor Hugo, Le Mans
  - Pôle Santé Sud, Le Mans
  - Centre Oscar Lambret, Lille
  - CHU de Lille, Lille
  - Centre Hospitalier Universitaire Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Centre Hopsitalier Lyon Sud, Lyon
  - Institut Paoli Calmettes, Marseille
  - AP-HM - Hôpital de la Timone, Marseille
  - CRLC Val d'Aurelle, Montpellier
  - Centre Hospitalier Universitaire Nice, Nice
  - Hopital Lariboisiere, Paris
  - Hopital Tenon, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Institut Curie, Paris
  - CHU - Hôpital de la Milétrie, Poitiers
  - Centre Hospitalier Universitaire Saint Etienne- Hopital Nord, Saint-Etienne
  - Ico-Centre Rene Gauducheau, Saint-Herblain
  - CHU Hautepierre, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Hospital Universitari Germans Trias I Pujol, Badalona, Spain

REFERENCES:
- [Result] Brigand C, Monneuse O, Mohamed F, Sayag-Beaujard AC, Isaac S, Gilly FN, Glehen O. Peritoneal mesothelioma treated by cytoreductive surgery and intraperitoneal hyperthermic chemotherapy: results of a prospective study. Ann Surg Oncol. 2006 Mar;13(3):405-12. doi: 10.1245/ASO.2006.05.041. Epub 2006 Jan 30. PMID 16485159
- [Result] Armstrong DK, Bundy B, Wenzel L, Huang HQ, Baergen R, Lele S, Copeland LJ, Walker JL, Burger RA; Gynecologic Oncology Group. Intraperitoneal cisplatin and paclitaxel in ovarian cancer. N Engl J Med. 2006 Jan 5;354(1):34-43. doi: 10.1056/NEJMoa052985. PMID 16394300
- [Derived] Classe JM, Meeus P, Hudry D, Wernert R, Quenet F, Marchal F, Houvenaeghel G, Bats AS, Lecuru F, Ferron G, Brigand C, Berton D, Gladieff L, Joly F, Ray-Coquard I, Durand-Fontanier S, Liberale G, Pocard M, Georgeac C, Gouy S, Guilloit JM, Guyon F, Costan C, Rousselet JM, de Guerke L, Bakrin N, Brument E, Martin E, Asselain B, Campion L, Glehen O; UNICANCER/CHIPOR Investigators. Hyperthermic intraperitoneal chemotherapy for recurrent ovarian cancer (CHIPOR): a randomised, open-label, phase 3 trial. Lancet Oncol. 2024 Dec;25(12):1551-1562. doi: 10.1016/S1470-2045(24)00531-X. Epub 2024 Nov 14. PMID 39549720